CLINICAL TRIAL: NCT01609257
Title: Phase 1-2, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Safety, Immunogenicity, and Efficacy Study in Healthy Adults of Intramuscular Norovirus Bivalent Virus-like Particle Vaccine in Experimental Human Norovirus GII.4 Disease
Brief Title: Norovirus Bivalent-Vaccine Efficacy Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LV03-105; U1111-1177-4095 (Registry Identifier: WHO)
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Prevention From Norovirus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norovirus Bivalent VLP Vaccine (Experimental): Norovirus Bivalent virus like particle (VLP) Vaccine (50 μg of GI.1 Norwalk VLP and 50 μg of GII.4 cVLP) adjuvanted with MPL and AI(OH)3, intramuscular (IM), Days 0 and 28.
  Interventions: Biological: Norovirus Bivalent Vaccine
- Placebo (Placebo Comparator): Saline Placebo (0.9% sodium chloride (NaCl) and preservative-free), intramuscular (IM), Days 0 and 28.
  Interventions: Biological: Saline Comparator

INTERVENTIONS:
Biological: Norovirus Bivalent Vaccine — 2 doses IM 28 days apart
  Arms: Norovirus Bivalent VLP Vaccine
Biological: Saline Comparator — 2 doses IM 28 days apart
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the norovirus vaccine is effective in preventing acute gastroenteritis due to the experimental human Norovirus GII.4 challenge dose. The purpose is also to evaluate the safety of the vaccine and the immunogenicity of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, a subject must meet the following criteria:

1. Signed informed consent.
2. Age 18 to 50 years (e.g., not reached their 50th birthday).
3. Good general health as determined by a screening evaluation within 45 days of randomization.
4. Expressed interest, availability, and understanding to fulfill the study requirements including measures to prevent Norovirus contamination of the environment and spread of infection and illness to the community. The prospective subjects must pass (≥70 % correct answers) a written examination on all aspects of the study before enrollment.
5. Available to return for follow-up visits following discharge from the inpatient unit and able to deliver stool specimens to the investigative site promptly with no plan to move within the duration of the study.
6. Female subjects must be of non-childbearing potential, or if of childbearing potential (as determined by the investigator) must be practicing abstinence or using an effective licensed method of birth control (e.g. oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device, or Depo-Provera; skin patch; vaginal ring or cervical cap) for 30 days prior to vaccination and must agree to continue such precautions during the study and for 60 days after the Challenge visit. Male subjects must agree not to father a child from the day of vaccination until 60 days after the Challenge visit.
7. Have a serum antibody titer of ≤1:1600 to the GII.4 Norovirus challenge strain as measured by Immunoglobulin G (IgG) P Particle Enzyme-Linked Immunosorbent Assay (ELISA.)
8. Demonstrated to be H Type 1 secretor positive by Histoblood Group Antigen (HBGA) binding assay of their saliva test. [This saliva test may be done at anytime prior to enrollment and does not need to be repeated.]
9. Negative serology for hepatitis C antibody, Human Immune Deficiency Virus (HIV) antibody, hepatitis B surface antigen, and Rapid Plasma Reagin (RPR).
10. Agrees not to participate in another clinical trial with an investigational product for the duration of the study (12 months after the last dose of study vaccine or placebo i.e. 393 days).

Exclusion Criteria:

To be eligible to participate in this study, a subject must NOT meet any of the following criteria:

1. Living with or having daily contact with children age 5 years or less or a woman known to be pregnant. This includes significant contact at home, school, day-care, or equivalent facilities.
2. Nursing mother.
3. Living with or having daily contact with childcare workers.
4. Living with or having daily contact with elderly persons aged 70 years or more, or infirmed, diapered individuals, persons with disabilities or incontinent persons. This includes work or visits to nursing homes and day-care or equivalent facilities.
5. History of any gastroenteritis suggestive of Norovirus illness since screening serum antibody IgG P Particle ELISA testing was done.
6. History of any gastroenteritis within the past 2 weeks.
7. History of chronic functional dyspepsia, chronic gastroesophageal reflux disease, peptic ulcer disease, gastrointestinal hemorrhage, gall bladder disease, inflammatory bowel disease, irritable bowel syndrome, frequent diarrhea, chronic constipation, malabsorption, maldigestion, major Gastrointestinal (GI) surgery, or diverticulitis anytime during the subject's lifetime or any other chronic GI disorders that would interfere with interpretation of symptoms or evaluation during the study.
8. Routine use of medication other than oral contraceptive agents, anti-hypertensives, anti-depressants, vitamins and minerals. The use of any other medications should be discussed with the Sponsor and/or Central Safety Monitor (CSM).
9. History of any of the following medical illnesses:

   * Immunosuppression (disease or treatments that may affect immune system function)
   * Diabetes (including gestational diabetes during the pregnancy that required treatment other than dietary).
   * Cancer (malignancy other than a resolved or excised skin lesion).
   * Heart disease (hospitalization for a heart attack, arrhythmia, or syncope)
   * Unconsciousness (other than a single brief "concussion")
   * Seizures (other than febrile seizures as a child <5 years old)
   * Asthma requiring treatment with inhaler or medication in the past 2 years.
   * Neuro-inflammatory disease
   * Autoimmune disease
   * Eating disorder
   * Chronic headaches associated with vomiting
   * Chronic vomiting syndrome
10. Any current illness requiring daily medication other than vitamins, minerals, birth control, anti-hypertensives or anti-depressants. The use of any other medications should be discussed with the Sponsor and/or CSM.
11. Allergies or hypersensitivity to any component of the vaccine or challenge virus.
12. Any clinically significant abnormality detected on physical examination, including:

    * Murmur (other than a functional, ie normal, murmur)
    * Focal neurological abnormality
    * Hepatosplenomegaly
    * Lymphadenopathy
    * Jaundice
13. Hypertension defined as BP > 150/90 mm Hg on two separate measurements. Chronic stable well-controlled hypertension on medications is allowed.
14. History of 3 or more hospitalizations for invasive bacterial infections (pneumonia, meningitis), acute or chronic dermatitis (e.g. eczema, seborrhea, psoriasis) or collagen vascular disease (e.g. Systemic Lupus Erythematosus (SLE) or dermatomyositis).
15. Presence of serious chronic illness.
16. Positive stool/fecal culture for bacterial pathogens (salmonella, campylobacter, E. coli 0157:H7, yersinia, or shigella) or positive stool/fecal screen for ova and parasites.
17. Employment in the food service industry, such as restaurants or cafeteria facilities. Specifically, this will include persons whose employment requires food processing in the 4 weeks following challenge.
18. Health-care workers with patient contact expected in the 4 weeks following challenge.
19. Expected contact (through employment or at home) with immunocompromised persons (HIV-positive, receiving immunosuppressive medications such as oral steroids or anti-neoplastic agents) in the 4 weeks following challenge.
20. Employment as an airline flight attendant scheduled to work in the 4 weeks following challenge.
21. Persons planning on taking a cruise in the 4 weeks following challenge.
22. Persons who plan to be living in a confined environment (e.g. ship, camp, or dormitory) within 4 weeks following challenge.
23. Persons who have consumed or plan to consume raw shellfish (e.g. oysters) from screening through post challenge Day 30.
24. Any of the following lab abnormalities (per the site local laboratory):

    * Absolute neutrophil count (ANC) outside the normal range
    * Total White Blood Cell Count (WBC) outside the normal range
    * Hemoglobin or hematocrit outside the normal range
    * Platelet count outside the normal range
    * Electrolytes [Sodium (Na), Potassium (K), Chloride (Cl), Carbon dioxide (CO2)], Blood Urea Nitrogen (BUN) and/or creatinine outside the normal range
    * Screening glucose > upper limit of normal (ULN). Fasting glucose is not required
    * Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), alkaline phosphatase, bilirubin (total and indirect), or Gamma Glutamyl Transferase (GGT) outside the upper limit of the normal range
    * Screening urinalysis with a value higher than "trace" positive for urine protein or urine glucose, or urine Red Blood Cells (RBCs) (≥3; other than women during menses).

    All of the above labs may be repeated if outside the normal limits. If repeated and continue outside site normal ranges, may enroll if determined by the Principal Investigator (PI) to be not clinically significant and discussed with the Sponsor and/or CSM.
25. For women of child bearing potential, positive serum pregnancy test within 14 days or positive urine pregnancy test within one day of randomization.
26. Temperature > 100.4°F orally, or symptoms of an acute self-limited illness such as an upper respiratory infection within 3 days of administering either dose of Norovirus Bivalent VLP vaccine or placebo control or the challenge product.
27. Resting heart rate >100 beats per minute or <55 beats per minute, respiratory rate ≥ 20 breaths per minute. If heart rate <55 beat per minute and the investigator determines that this is not clinically significant and heart rate increases > 55 beats per minute on moderate exercise, subject will not be excluded. Vital signs may be repeated.
28. Clinically abnormal screening electrocardiogram (ECG) defined as pathologic Q waves and significant ST-T wave changes; criteria for left ventricular hypertrophy; and any non-sinus rhythm excluding isolated premature atrial contractions.
29. Previous participation in a study of experimental norovirus infection or norovirus vaccine.
30. Study site personnel or their family members
31. Significant history of psychiatric hospitalization, alcohol abuse, or illicit drug use.
32. Receipt of a licensed live vaccine within 28 days or a licensed inactivated vaccine within 14 days of administration of either dose of vaccine or placebo or the challenge product.
33. Completion of an investigational vaccine or drug study within 7 days of randomization.
34. Receipt of systemic corticosteroids for greater than 7 days within the past six months.
35. Regular use of laxatives or anti-motility agents.
36. Receipt of blood or blood products within the past six months.
37. Subjects who are unwilling or unable to cease smoking from entry to the inpatient facility until discharge from the inpatient facility.
38. Other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a subject participating in the trial, would render the subject unable to comply with the protocol, or would interfere with the evaluation of the Vaccination stage or the evaluation of the Challenge stage.

Challenge Stage Exclusion Criteria

The following additional exclusion criteria must not be met prior to admission to the inpatient unit for Challenge:

1. Use of antibiotics within the 7 days prior to entry into the inpatient challenge facility.
2. Use of any H-2 receptor antagonists (e.g. Tagamet, Zantac, and Pepcid), proton pump inhibitors (e.g. Prilosec, Protonix, and Prevacid), or prescription acid suppression medication or over the counter antacids within 72 hours of the challenge.
3. Use of prescription or Over the Counter (OTC) medications containing acetaminophen, aspirin, ibuprofen, and/or other non-steroidal anti-inflammatory drugs within 48 hours prior to challenge.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bernstein, MD, Principal Investigator — Cincinatti Children's Hospital; Mohamed S Al-Ibrahim, MB, ChB, Principal Investigator — SNBL Clinical Pharmacology Center; David Y Graham, MD, Principal Investigator — Baylor College of Medicine; Robert L Atmar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; G. Marshall Lyon, MD, Principal Investigator — Emory University; John J Treanor, MD, Principal Investigator — University of Rochester
Locations (5):
- United States (5):
  - Emory University, Atlanta, Georgia
  - SNBL, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Bernstein DI, Atmar RL, Lyon GM, Treanor JJ, Chen WH, Jiang X, Vinje J, Gregoricus N, Frenck RW Jr, Moe CL, Al-Ibrahim MS, Barrett J, Ferreira J, Estes MK, Graham DY, Goodwin R, Borkowski A, Clemens R, Mendelman PM. Norovirus vaccine against experimental human GII.4 virus illness: a challenge study in healthy adults. J Infect Dis. 2015 Mar 15;211(6):870-8. doi: 10.1093/infdis/jiu497. Epub 2014 Sep 9. PMID 25210140
- [Derived] Atmar RL, Bernstein DI, Lyon GM, Treanor JJ, Al-Ibrahim MS, Graham DY, Vinje J, Jiang X, Gregoricus N, Frenck RW, Moe CL, Chen WH, Ferreira J, Barrett J, Opekun AR, Estes MK, Borkowski A, Baehner F, Goodwin R, Edmonds A, Mendelman PM. Serological Correlates of Protection against a GII.4 Norovirus. Clin Vaccine Immunol. 2015 Aug;22(8):923-9. doi: 10.1128/CVI.00196-15. Epub 2015 Jun 3. PMID 26041041
- [Derived] Sundararajan A, Sangster MY, Frey S, Atmar RL, Chen WH, Ferreira J, Bargatze R, Mendelman PM, Treanor JJ, Topham DJ. Robust mucosal-homing antibody-secreting B cell responses induced by intramuscular administration of adjuvanted bivalent human norovirus-like particle vaccine. Vaccine. 2015 Jan 15;33(4):568-76. doi: 10.1016/j.vaccine.2014.09.073. Epub 2014 Nov 22. PMID 25444793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 16 June 2012 to 18 March 2014.
Pre-assignment Details: Healthy Volunteers were enrolled equally in 1 of 2 treatment groups, Norovirus Bivalent VLP Vaccine or Placebo.
Groups:
- Placebo: Saline (0.9% NaCl and preservative-free), IM, Days 0 and 28.
Period: Overall Study
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Started | 67 | 65
Received 2 Doses | 63 | 64
Received Challenge Product | 56 | 53
Completed | 61 | 57
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Voluntary Withdrawal by Subject | 0 | 1
Not completed — Non-compliance/Protocol deviation | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo | Total
Number analyzed (Participants) | 67 | 65 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.2) | 32.1 (9.3) | 32.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 35 | 33 | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic | 65 | 63 | 128
  Hispanic | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Black/African American | 37 | 36 | 73
  White | 25 | 26 | 51
  Multi-Racial | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 67 | 65 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Viral AGE Clinical Illness and Fecal Virus Excretion Detected by RT-PCR OR 4-Fold Rise In Anti-GII.4 Norovirus P Particle Antibody Titer
Description: Viral AGE due to Norovirus GII.4 strain during the inpatient stay that meets clinical illness definition 1,2 or 3 and positive for infection as measured by fecal virus excretion detected by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) OR a 4-fold rise in Immunoglobulin G Enzyme-Linked Immunosorbent Assay (IgG ELISA) anti-GII.4 norovirus P particle antibody titer from pre-challenge (Within 2 weeks of Challenge Day 0) to post-challenge (Challenge Day 30). The clinical illness definitions are 1: diarrhea (defined as ≥ 3 loose or liquid stools OR >400-600 grams of loose or liquid stools produced in any 24-hour period), 2: vomiting (defined as ≥ 2 vomiting episodes in any 24-hour period) or 3. One Vomiting episode plus any loose or liquid stool in any 24-hour period OR one vomiting episode plus at least 2 of the following 5 events: nausea, fever ≥99.7°F orally, abdominal cramps or pains, abdominal gurgling or bloating, or myalgia in any 24-hour period.
Time Frame: Symptoms collected from Challenge dose (at least 28 days after dose 2) to discharge (at least 96 hours after challenge dose)
Population: Modified intent-to-treat population (mITT) included all participants who received at least one dose of study drug, challenge stage.
Measure: Number; unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 56 | 53
percentage of participants | 26.8 | 32.1
Statistical Analysis 1: Comparison: Norovirus Bivalent VLP Vaccine vs Placebo; Test type: Superiority or Other; p = 0.674, Fisher Exact — No multiplicity adjustment

2. Primary Outcome: Percentage of Participants Experiencing Solicited Local Adverse Events Within 7 Days Post-Dose 1
Description: Local Adverse Events included local injection site reactions/symptoms: pain, tenderness, redness, and swelling.
Time Frame: Within 7 days post-dose 1
Population: MITT population included all participants who received at least one dose of study drug. Data is missing for 2 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 66 | 64
percentage of participants | 66.7 [54.0 to 77.8] | 28.1 [17.6 to 40.8]

3. Primary Outcome: Percentage of Participants Experiencing Solicited Local Adverse Events Within 7 Days Post-Dose 2
Description: Local Adverse Events included local injection site reactions/symptoms: pain, tenderness, redness, and swelling.
Time Frame: Within 7 days post-dose 2
Population: Participants from the MITT population, all participants who received at least one dose of study drug, who received a second dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants | 54.0 [40.9 to 66.6] | 20.6 [11.5 to 32.7]

4. Primary Outcome: Percentage of Participants Experiencing Solicited Systemic Adverse Events Within 7 Days Post-Dose 1
Description: Systemic signs or symptoms included: elevated daily oral temperature (fever), headache, fatigue, muscle aches, chills, joint aches and gastrointestinal symptoms of nausea, vomiting, diarrhea, abdominal cramps/pain.
Time Frame: Within 7 days post-dose 1
Population: MITT included all participants who received at least one dose of study drug. Data is missing for 2 participants.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 66 | 64
percentage of particpants | 36.4 [24.9 to 49.1] | 32.8 [21.6 to 45.7]

5. Primary Outcome: Percentage of Participants Experiencing Solicited Systemic Adverse Events Within 7 Days Post-Dose 2
Description: Systemic signs or symptoms included: elevated fever, headache, fatigue, muscle aches, chills, joint aches and gastrointestinal symptoms of nausea, vomiting, diarrhea, abdominal cramps/pain.
Time Frame: Within 7 days post-dose 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of particpants | 30.2 [19.2 to 43.0] | 19.0 [10.2 to 30.9]

6. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) 365 Days Following the Last Study Vaccination
Description: A SAE was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: 365 Days Following Dose 2 (Up to 393 days)
Population: MITT population included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
percentage of participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With 4-Fold Rise In Serum P-Particle Antibody Titer by ELISA or Detection of Norovirus GII.4 by RT-PCR in the Stool
Time Frame: Pre Challenge to 30 Days Post Challenge
Population: MITT population included all participants who received at least one dose of study drug, Challenge stage.
Measure: Number; unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 56 | 53
percentage of participants
  RT-PCR Alone | 53.6 | 60.4
  4-Fold rise in P-particle ELISA alone; n=56,51 | 7.1 | 52.9
  Either RT-PCR or 4-fold rise in P-particle;n=56,52 | 53.6 | 61.5

8. Secondary Outcome: Severity of Viral AGE Due to GII.4 Strain Assessed by Modified Vesikari Scoring System During the Inpatient Phase
Description: Vesikari Scoring System assesses the following symptoms: duration of diarrhea (days), maximum number of diarrheal stools/24 hours, duration of vomiting (days), maximum number of vomiting episodes/24 hours, fever and dehydration. Since the typical inpatient phase was four days in length, the duration of diarrhea scoring was modified to fit this time frame. Modified Vesikari Scale Total Score=0 to 17. Higher numbers are worse.
Time Frame: as for outcome 1
Population: Participants from the MITT population, all participants who received at least one dose of study drug, challenge stage with Viral AGE.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 15 | 17
score on a scale | 4.4 (2.0) | 7.1 (2.1)
Statistical Analysis 1: Comparison: Norovirus Bivalent VLP Vaccine vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — Statistically significant at p<0.05. No multiplicity adjustment

9. Secondary Outcome: Severity of Viral AGE Due to GII.4 Strain Assessed by Post-Challenge Symptom Collection During the Inpatient Phase
Description: Score 1 was based on a subset of symptoms including: elevated oral temperature, myalgia, nausea, abdominal cramps, bloating, diarrhea, and vomiting. Score 2 was based on all Score 1 symptoms plus fatigue/malaise, chills, and loss of appetite. Total Score 1=0 to 20 and Total Score 2=0 to 29. Higher numbers are worse.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 15 | 17
score on a scale
  Score 1 | 1.8 (1.0) | 3.3 (2.0)
  Score 2 | 2.7 (1.5) | 4.5 (3.0)
Statistical Analysis 1: Comparison: Norovirus Bivalent VLP Vaccine vs Placebo; Score 1; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — Statistically significant at p<0.05. No multiplicity adjustment
Statistical Analysis 2: Comparison: Norovirus Bivalent VLP Vaccine vs Placebo; Score 2; Test type: Superiority or Other; p = 0.037, Wilcoxon (Mann-Whitney) — Statistically significant at p<0.05. No multiplicity adjustment

10. Secondary Outcome: Duration of Viral AGE Due to GII.4 Strain During the Inpatient Phase
Description: Duration of symptoms was determined by a blinded committee review of each participant's symptoms.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 15 | 17
hours | 32.1 [10.4 to 60.0] | 38.0 [2.0 to 71.0]
Statistical Analysis 1: Comparison: Norovirus Bivalent VLP Vaccine vs Placebo; Test type: Superiority or Other; p = 0.199, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Percentage of Participants With GII.4 Norovirus Positive RT-PCR in the Stool During the Inpatient and /or Outpatient Phase
Time Frame: Pre Challenge to 30 Days Post Challenge
Population: Participants from the MITT population, all participants with at least one dose of study drug, challenge stage with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 56 | 53
percentage of participants
  Pre-Challenge | 0.0 | 0.0
  Day 1 (n=54,53) | 1.9 | 3.8
  Day 2 (n=52,52) | 38.5 | 30.8
  Day 3 (n=55,51) | 45.5 | 51.0
  Day 4 (n=52,47) | 44.2 | 55.3
  Day 10 (n=55,51) | 21.8 | 33.3
  Day 30 (n=56,52) | 0.0 | 0.0
  Any Day 1 to 30 | 53.6 | 60.4
Statistical Analysis 1: Comparison: Norovirus Bivalent VLP Vaccine vs Placebo; Any Day 1 to 30; Test type: Superiority or Other; p = 0.562, Fisher Exact — Comparison of % Positive

12. Secondary Outcome: Percentage of Participants With GII.4 Seroresponse Rate (4-fold Rise) From Pre-challenge Day 0 to Post-Challenge Day 30
Description: Seroresponse was a 4-fold increase in IgG ELISA anti-GII.4 norovirus P particle antibody titer from pre-challenge to post-challenge.
Time Frame: Pre Challenge to 30 Days Post Challenge
Population: Participants from the MITT population, all participants who received at least one dose of study drug, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 56 | 51
percentage of participants | 7.1 [2.0 to 17.3] | 52.9 [38.5 to 67.1]

13. Other Pre Specified Outcome: Correlation of GII.4 Serum HBGA Antibodies Prior to Challenge Associated With Protection From GII.4 Illness
Description: Percentage of placebo subjects HBGA seropositive pre-challenge by illness status.
Time Frame: Pre Challenge to Day 30 Post Challenge
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Groups:
- Placebo_Not Ill: Saline (0.9% NaCl and preservative-free), IM, Days 0 and 28.
Arm/Group | Placebo | Placebo_Not Ill
Number analyzed (Participants) | 16 | 36
percentage of participants | 6.3 | 47.2

14. Other Pre Specified Outcome: Correlation of GII.4 Serum HGBA Antibodies Prior to Challenge Associated With Protection From GII.4 Infection
Description: Percentage of placebo subjects HBGA seropositive pre-challenge by infection status.
Time Frame: Pre Challenge to Day 30 Post Challenge
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Groups:
- Placebo_Not Infected: Saline (0.9% NaCl and preservative-free), IM, Days 0 and 28.
Arm/Group | Placebo | Placebo_Not Infected
Number analyzed (Participants) | 31 | 20
percentage of participants | 12.9 | 65.0

15. Secondary Outcome: Pan-Ig ELISA - Anti-Norovirus GI.1 VLP Geometric Mean Fold Rise (GMFR) From Baseline
Time Frame: Baseline to 28 days Post Dose 1 and 28 days Post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
ratio
  28 days Post Dose 1 (n=63, 63) | 65.4 [47 to 91] | 1.0 [0.9 to 1.1]
  28 days Post Dose 2 (n= 61, 58) | 61.2 [43.9 to 85.2] | 0.9 [0.8 to 1.0]

16. Secondary Outcome: Percentage of Participants With Pan-Ig ELISA - Anti-Norovirus GI.1 VLP Seroresponse (4-fold Rise) From Baseline
Time Frame: Baseline, 28 days Post Dose 1 and 28 days Post Dose 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants
  28 days Post Dose 1 (n=63, 63) | 100.0 [94.3 to 100.0] | 1.6 [0.0 to 8.5]
  28 days Post Dose 2 (n= 61, 58) | 100.0 [94.1 to 100.0] | 3.4 [0.4 to 11.9]

17. Secondary Outcome: Pan-Ig ELISA - Anti-Norovirus GI.1 VLP Geometric Mean Titer (GMT)
Time Frame: Baseline, 28 days Post Dose 1 and 28 days Post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
titer
  Baseline (Pre-Dose 1) | 1857.6 [1314.1 to 2626.0] | 1671.1 [1188.9 to 2348.7]
  28 days Post Dose 1 (n=63, 63) | 127209.7 [99321.5 to 162928.4] | 1577.6 [1105.5 to 2251.3]
  28 days Post Dose 2 (n=61, 58) | 120552.8 [98844.3 to 147029.0] | 1606.3 [1097.7 to 2350.6]

18. Secondary Outcome: Pan-Ig ELISA - Anti-Norovirus GII.4 cVLP GMFR From Baseline
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
ratio
  28 days Post Dose 1 (n=63, 63) | 12.2 [8.3 to 17.9] | 1.0 [0.9 to 1.1]
  28 days Post Dose 2 (n=61, 58) | 10.4 [7.5 to 14.5] | 1.1 [0.9 to 1.3]

19. Secondary Outcome: Percentage of Participants With Pan-Ig ELISA - Anti-Norovirus GII.4 cVLP Seroresponse From Baseline
Description: Seroresponse was defined as a 4-Fold Rise from Baseline.
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants
  28 days Post Dose 1 (n=63, 63) | 82.5 [70.9 to 90.9] | 1.6 [0.0 to 8.5]
  28 days Post Dose 2 (n=61, 58) | 88.5 [77.8 to 95.3] | 1.7 [0.0 to 9.2]

20. Secondary Outcome: Pan-Ig ELISA - Anti-Norovirus GII.4 cVLP GMT
Time Frame: Baseline, 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
titer
  Baseline (Pre-Dose 1) | 5120.0 [3754.9 to 6981.3] | 4958.8 [3776.8 to 6510.8]
  28 days Post Dose 1 (n=63, 63) | 63604.8 [49961.2 to 80974.3] | 4845.9 [3640.0 to 6451.4]
  28 days Post Dose 2 (n=61, 58) | 56303.8 [45918.6 to 69037.7] | 5306.9 [3822.1 to 7368.5]

21. Secondary Outcome: ELISA Immunoglobulin A (IgA)- Anti-Norovirus GI.1 VLP Geometric Mean Fold Rise (GMFR) From Baseline
Time Frame: Baseline to 28 days Post Dose 1 and 28 days Post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
ratio
  28 days Post Dose 1 (n=63, 63) | 16.3 [11.5 to 23.2] | 1.0 [1.0 to 1.1]
  28 days Post Dose 2 (n= 61, 58) | 11.5 [8.2 to 16.2] | 1.0 [1.0 to 1.1]

22. Secondary Outcome: Percentage of Participants With ELISA IgA- Anti-Norovirus GI.1 VLP Seroresponse (4-fold Rise) From Baseline
Time Frame: Baseline to 28 days Post Dose 1 and 28 days Post Dose 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants
  28 days Post Dose 1 (n=63, 63) | 85.7 [74.6 to 93.3] | 0.0 [0.0 to 5.7]
  28 days Post Dose 2 (n= 61, 58) | 80.3 [68.2 to 89.4] | 0.0 [0.0 to 6.2]

23. Secondary Outcome: ELISA IgA- Anti-Norovirus GI.1 VLP Geometric Mean Titer (GMT)
Time Frame: Baseline, 28 days Post Dose 1 and 28 days Post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
titer
  Baseline (Pre-Dose 1) | 4.1 [3.5 to 4.8] | 4.0 [3.5 to 4.5]
  28 days Post Dose 1 (n=63, 63) | 66.9 [46.8 to 95.7] | 4.0 [3.5 to 4.7]
  28 days Post Dose 2 (n=61, 58) | 47.5 [33.2 to 67.8] | 4.0 [3.5 to 4.7]

24. Secondary Outcome: ELISA IgA- Anti-Norovirus GII.4 cVLP GMFR From Baseline
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
ratio
  28 days Post Dose 1 (n=63, 63) | 9.0 [6.7 to 12.1] | 1.0 [0.9 to 1.1]
  28 days Post Dose 2 (n=61, 58) | 7.7 [6.0 to 9.9] | 1.1 [0.9 to 1.2]

25. Secondary Outcome: Percentage of Participant With ELISA IgA- Anti-Norovirus GII.4 cVLP Seroresponse From Baseline
Description: Seroresponse was defined as a 4-Fold Rise from Baseline.
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants
  28 days Post Dose 1 (n=63, 63) | 73.0 [60.3 to 83.4] | 3.2 [0.4 to 11.0]
  28 days Post Dose 2 (n=61, 58) | 72.1 [59.2 to 82.9] | 1.7 [0.0 to 9.2]

26. Secondary Outcome: ELISA IgA- Anti-Norovirus GII.4 cVLP GMT
Time Frame: Baseline, 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
titer
  Baseline (Pre-Dose 1) | 5.9 [4.8 to 7.4] | 5.8 [4.8 to 7.1]
  28 days Post Dose 1 (n=63, 63) | 54.1 [43.3 to 67.6] | 6.1 [5.0 to 7.4]
  28 days Post Dose 2 (n=61, 58) | 47.0 [39.1 to 56.5] | 6.2 [5.0 to 7.7]

27. Secondary Outcome: HBGA (PGM) - Anti-Norovirus GI.1 VLP GMFR From Baseline
Description: HBGA (PGM) is Histoblood Group Antigen (Pig Gastric Mucin).
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
ratio
  28 days Post Dose 1 (n=63, 63) | 25.6 [19.1 to 34.3] | 1.0 [0.9 to 1.1]
  28 days Post Dose 2 (n=61, 58) | 31.8 [25.8 to 39.1] | 1.0 [0.9 to 1.1]

28. Secondary Outcome: Percentage of Participants With HBGA (PGM) - Anti-Norovirus GI.1 VLP Seroresponse From Baseline
Description: Seroresponse was defined as a 4-Fold Rise from Baseline
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants
  28 days Post Dose 1 (n=63, 63) | 95.2 [86.7 to 99.0] | 0.0 [0.0 to 5.7]
  28 days Post Dose 2 (n=61, 58) | 100.0 [94.1 to 100.0] | 0.0 [0.0 to 6.2]

29. Secondary Outcome: HBGA (PGM) - Anti-Norovirus GI.1 VLP GMT
Time Frame: Baseline, 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
titer
  Baseline (Pre-Dose 1) | 17.5 [14.6 to 20.9] | 15.2 [13.2 to 17.5]
  28 days Post Dose 1 (n=63, 63) | 456.2 [324.4 to 641.6] | 15.4 [13.5 to 17.6]
  28 days Post Dose 2 (n=61, 58) | 573.5 [453.0 to 726.1] | 15.1 [13.1 to 17.4]

30. Secondary Outcome: HBGA (PGM) - Anti-Norovirus GII.4 cVLP GMFR From Baseline
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
ratio
  28 days Post Dose 1 (n=63, 63) | 8.0 [6.2 to 10.3] | 1.0 [0.9 to 1.0]
  28 days Post Dose 2 (n=61, 58) | 6.6 [5.3 to 8.1] | 1.0 [0.9 to 1.2]

31. Secondary Outcome: Percentage of Participants With HBGA (PGM) - Anti-Norovirus GII.4 cVLP Seroresponse From Baseline
Description: Seroresponse was defined as a 4-Fold Rise from Baseline.
Time Frame: Baseline to 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 63 | 63
percentage of participants
  28 days Post Dose 1 (n=63, 63) | 69.8 [57.0 to 80.8] | 0.0 [0.0 to 5.7]
  28 days Post Dose 2 (n=61, 58) | 73.8 [60.9 to 84.2] | 1.7 [0.0 to 9.2]

32. Secondary Outcome: HBGA (PGM) - Anti-Norovirus GII.4 cVLP GMT
Time Frame: Baseline, 28 days post Dose 1 and 28 days post Dose 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
titer
  Baseline (Pre-Dose 1) | 119.2 [104.8 to 135.5] | 127.5 [109.5 to 148.5]
  28 days Post Dose 1 (n=63, 63) | 971.5 [794.2 to 1188.3] | 126.4 [107.7 to 148.2]
  28 days Post Dose 2 (n=61, 58) | 803.0 [679.8 to 948.7] | 136.7 [113.3 to 165.0]

33. Secondary Outcome: Percentage of Participants With Unsolicited Non-Serious [i.e Other Than SAEs] Adverse Events (AEs)
Description: Unsolicited AEs indicates any and all AEs that occurred other than those that were solicited.
Time Frame: Vaccination Stage: Initial vaccination until 28 days after second vaccination; or Challenge Stage: the day of challenge until 60 days after challenge
Population: MITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Number analyzed (Participants) | 67 | 65
percentage of participants
  Post Dose 1 | 10.4 [4.3 to 20.3] | 23.1 [13.5 to 35.2]
  Post Dose 2 (n=63, 64) | 14.3 [6.7 to 25.4] | 18.8 [10.1 to 30.5]
  Challenge Stage | 39.3 [26.5 to 53.2] | 50.9 [36.8 to 64.9]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 393 Days. Non-Serious Unsolicited Events Post Vaccination: Initial vaccination until 28 days after second vaccination
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Norovirus Bivalent VLP Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/65
Other Adverse Events (participants affected / at risk) | 10/67 | 7/65
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Norovirus Bivalent VLP Vaccine (N=67) | Placebo (N=65)
Nasopharyngitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Blood glucose increased (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.